CLINICAL TRIAL: NCT04210063
Title: Effect of Inspiratory Muscle Training (IMT) on Breathing, Balance, and Blood Pressure Maintenance in Spinal Cord Injury (SCI)
Brief Title: Orthostatic, Respiratory, Balance-Intervention
Acronym: ORB-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Foundation for Physical Therapy, Inc. (Industry); The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Lawrence Cahalin, Clinical Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190838
Record Dates: First submitted 2019-12-18; First posted 2019-12-24 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Spinal Cord Injuries
Keywords: Breathing; Diaphragm; Balance; Blood Pressure
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMT Intervention (Experimental): During the first month, participants will be in a month-long control wash in period where no intervention will be provided. During the second month, participants will be in a 4-week daily IMT intervention period. During the third month, participants will be in a month-long efficacy period with no intervention provided.
  Interventions: Other: Inspiratory Muscle Training (IMT)

INTERVENTIONS:
Other: Inspiratory Muscle Training (IMT) — IMT is a breathing training technique customized to participant's breathing capacity. Using a handheld electronic manometer (Pro2Fit from Smithfield), a study personnel will initiate training at 40-60% maximal inspiratory pressure. Adjustments will be customized to where the participant reports a difficulty of training between 4-6 out of 10. Training sessions will be performed about 30 minutes a day for 28 consecutive days.

SUMMARY:
The purpose of this study is to help understand how training breathing muscles will impact balance, blood pressure, and quality of life of participants with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Upper/lower/both extremity weakness or paralysis resulting from SCI with ASIA Impairment Scale (AIS) grades A-C who use a wheelchair as primary means of mobility.
2. ≥1 year post-injury
3. Willingness to participate in the study and provide consent.

Exclusion Criteria:

1. Inability to understand the consent form or consent process
2. Reliance on a mechanical ventilator.
3. Use of Betablockers
4. Inability to travel to The Miami Project for weekly sessions during intervention month
5. Any complication that would limit transfer ability, or compromise supine or sitting tolerance, including but not limited to:

   * Fracture, dislocation, or malformations affecting supine or sitting tolerance.
   * Spinal instability.
   * Pressure ulcers or skin integrity issues on contact surfaces that would prohibit sitting or lying in supine.
6. Individuals who are able to stand independently or with a walker
7. Unresolved deep vein thrombosis (DVT).
8. Hospitalization due to autonomic dysreflexia in the last 3 months.
9. Pregnancy determined by urine testing in sexually active females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Percent Compliance of Training Sessions | 4 weeks
  Feasibility of the IMT protocol will be reported as the percentage of completed daily sessions out of the 28 total session days.
Percent Compliance of Training Minutes | 4 weeks
  Feasibility of the IMT protocol will also be reported as the percentage of completed total time out of the 840 minutes total expected session minutes(30 minutes daily for 28 days).
Maximal Inspiratory Pressure (MIP) | Week 12
  MIP measured in cm H2O will be assessed using the Pro2 handheld inspiratory measurement and training device connected to a tablet, phone or desktop
Sustained Maximal Inspiratory Pressure (SMIP) | Week 12
  SMIP measured in pressure-time units (PTU) will be assessed using the Pro2 handheld inspiratory measurement and training device connected to a tablet, phone or desktop.
Standard deviation of normal R-R intervals (SDNN) | Week 12
  SDNN, measured in milliseconds, will be derived from signals obtained by a Polar monitor (with elastic chest strap sensor) and analyzed using Kubios Heart Rate Variability (HRV) Analysis Software.
Root Mean Squared of Successive Differences between Normal Heartbeats (rMSSD) | Week 12
  rMSSD, measured in milliseconds, will be derived from signals obtained by a Polar monitor (with elastic chest strap sensor) and analyzed using Kubios Heart Rate Variability (HRV) Analysis Software.
Systolic Blood Pressure (SBP) | Week 12
  Brachial systolic BP, evaluated in mmHg, will be evaluated using the contralateral arm with a Spot Vitals Monitor.
Functional Seated Balance | Week 12
  Functional Seated Balance will be measured using the Function in Sitting Test for SCI (FIST-SCI). FIST-SCI consist of 14 different standardized seated balance tasks and scored on a 5-point ordinal scale from 0-4. A higher score indicates increased independence.
Quality of Life (QoL) | Week 12
  QoL will be measured using the Quality of Life Index, SCI version (QOLI-SCI). QOLI-SCI is a set of two 37-items questionnaire with total scores ranging from 74 to 444 with the higher score indicating increased quality of life.
Independence | Week 12
  Independence will be measured using the Spinal Cord Independence Measured (SCIM). SCIM has a total score ranging from 0-100 with the higher score indicating increased independence.

SECONDARY OUTCOMES:
Inspiratory Duration (ID) | Week 12
  ID measured in seconds will be assessed using the Pro2 handheld inspiratory measurement and training device connected to a tablet, phone or desktop.
Forced Vital Capacity | Week 12
  FVC, evaluated in liters, will be measured using a handheld digital spirometer device.
Forced Expiratory Volume in one Second (FEV1) | Week 12
  FEV1, evaluated in liters, will be measured using a handheld digital spirometer device.
Peak Expiratory Flow (PEF) | Week 12
  PEF, evaluated in liters/minute, will be measured using a handheld digital spirometer device.
Maximal Expiratory Pressure (MEP) | Week 12
  MEP, evaluated in cm H2O, will be measured using a handheld digital spirometer device.
Heart Rate Variability (HRV) Frequency | Week 12
  Low Frequency (LF) and High Frequency (HF) Power, reported in percentage, will be derived from signals obtained by a Polar monitor (with elastic chest strap sensor) and analyzed using Kubios Heart Rate Variability (HRV) Analysis Software.
Diastolic Blood Pressure (DBP) | Week 12
  Brachial diastolic BP, evaluated in mmHg, will be evaluated using the contralateral arm with a Spot Vitals Monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Cahalin, PhD, Principal Investigator — University of Maimi
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDonald T, Stiller K. Inspiratory muscle training is feasible and safe for patients with acute spinal cord injury. J Spinal Cord Med. 2019 Mar;42(2):220-227. doi: 10.1080/10790268.2018.1432307. Epub 2018 Feb 5. PMID 29400990
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Aslan SC, Randall DC, Krassioukov AV, Phillips A, Ovechkin AV. Respiratory Training Improves Blood Pressure Regulation in Individuals With Chronic Spinal Cord Injury. Arch Phys Med Rehabil. 2016 Jun;97(6):964-73. doi: 10.1016/j.apmr.2015.11.018. Epub 2015 Dec 21. PMID 26718236
- [Background] Mello PR, Guerra GM, Borile S, Rondon MU, Alves MJ, Negrao CE, Dal Lago P, Mostarda C, Irigoyen MC, Consolim-Colombo FM. Inspiratory muscle training reduces sympathetic nervous activity and improves inspiratory muscle weakness and quality of life in patients with chronic heart failure: a clinical trial. J Cardiopulm Rehabil Prev. 2012 Sep-Oct;32(5):255-61. doi: 10.1097/HCR.0b013e31825828da. PMID 22785143
- [Background] Anderson KD, Acuff ME, Arp BG, Backus D, Chun S, Fisher K, Fjerstad JE, Graves DE, Greenwald K, Groah SL, Harkema SJ, Horton JA 3rd, Huang MN, Jennings M, Kelley KS, Kessler SM, Kirshblum S, Koltenuk S, Linke M, Ljungberg I, Nagy J, Nicolini L, Roach MJ, Salles S, Scelza WM, Read MS, Reeves RK, Scott MD, Tansey KE, Theis JL, Tolfo CZ, Whitney M, Williams CD, Winter CM, Zanca JM. United States (US) multi-center study to assess the validity and reliability of the Spinal Cord Independence Measure (SCIM III). Spinal Cord. 2011 Aug;49(8):880-5. doi: 10.1038/sc.2011.20. Epub 2011 Mar 29. PMID 21445081
- [Background] Janssens L, McConnell AK, Pijnenburg M, Claeys K, Goossens N, Lysens R, Troosters T, Brumagne S. Inspiratory muscle training affects proprioceptive use and low back pain. Med Sci Sports Exerc. 2015 Jan;47(1):12-9. doi: 10.1249/MSS.0000000000000385. PMID 24870567
- [Background] May LA, Warren S. Measuring quality of life of persons with spinal cord injury: external and structural validity. Spinal Cord. 2002 Jul;40(7):341-50. doi: 10.1038/sj.sc.3101311. PMID 12080462
- [Derived] Palermo AE, Nash MS, Kirk-Sanchez NJ, Cahalin LP. Adherence to and impact of home-based high-intensity IMT in people with spinal cord injury: a pilot study. Spinal Cord Ser Cases. 2022 Oct 30;8(1):85. doi: 10.1038/s41394-022-00551-5. PMID 36309488